CLINICAL TRIAL: NCT04657939
Title: Targeting Beta-cell Failure in Lean Patients With Type 2 Diabetes
Acronym: Lean-DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Eylem Levelt, Principal Investigator, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 265208; 18/0005908 (Other Grant/Funding Number: Diabetes UK); 19/WM/0365 (Other: West Midlands- Black Country Research Ethics Committee)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liraglutide-Pioglitazone (Active Comparator): Participants randomised to receive liraglutide treatment for 16 weeks, followed by an 8 week washout then commencing 16 weeks of treatment with pioglitazone.
  Interventions: Drug: Liraglutide; Drug: Pioglitazone
- Pioglitazone-Liraglutide (Active Comparator): Participants randomised to receive pioglitazone treatment for 16 weeks, followed by an 8 week washout then commencing 16 weeks of treatment with liraglutide.
  Interventions: Drug: Liraglutide; Drug: Pioglitazone

INTERVENTIONS:
Drug: Liraglutide — Liraglutide 0.6mg once daily by subcutaneous injection escalated to 1.2mg after 2 weeks.
Drug: Pioglitazone — Pioglitazone 15mg once daily tablets taken orally escalated to 30mg after 2 weeks then escalated to 45mg after another 2 weeks.

SUMMARY:
The majority of people with type 2 diabetes (T2D) are overweight, and while weight gain is a major contributor to diabetes, a minority of patients with T2D are not overweight or obese. The reasons why lean or normal body weight individuals develop T2D (lean-T2D) are not yet understood. T2D occurs when the body does not produce enough insulin, or becomes less sensitive to its effects. Insulin acts like a key to allow sugar into cells and if someone is overweight that key works less well. Recent research suggests that T2D in lean people should be considered a different disease from the diabetes associated with obesity and the main problem in lean-T2D patients may be a reduced capacity of insulin secretion. However, some researchers argue that many seemingly thin people carry more fat than muscle, making them trim on the outside, but fat on the inside, and they are in fact not truly lean. This implies that just like overweight diabetics, lean diabetics also have high resistance to insulin. The main aim of this research is to better understand the main driver of T2D in lean individuals, as this will determine how best to treat these individuals.

There are many different types of drugs for treating T2D. Liraglutide improves insulin secretion capacity of the pancreas. Pioglitazone reduces resistance to insulin action. The investigators will compare the actions of these diabetes drugs on the blood supply and the heart's energy levels in lean-T2D and obese-T2D patients. This will allow the investigators to determine the ideal treatment strategies for improving cardiovascular health in lean-T2D patients, and better understand the role of impaired insulin secretory capacity, insulin resistance and excess fat deposition specifically in this group.

DETAILED DESCRIPTION:
This is a single centre, open-label, randomized, cross-over study. Participants will attend 4 visits in total over the course of approximately 40 weeks. Two cohorts of patients will be recruited: 28 lean-T2D patients and 28 obese-T2D patients.

Potential participants will be invited to the research centre for a screening/ baseline visit (Visit 1). At this visit, the participants will be given the Participant Information Sheet (PIS) to read through, and given the opportunity to ask questions. If they are interested in participating, their consent will be taken in written form. Each participant will then have a series of non-invasive tests. At this baseline visit, the following assessments will be done:

* Review of medical history and concomitant medications;
* Review of history of diabetes and complications;
* Review of inclusion/exclusion criteria;
* Collection of demographic data;
* Vital signs;
* Physical examination;
* Height and weight;
* Blood pressure;
* Urine pregnancy test in women of childbearing potential;
* Venepuncture (fasting sample): 20mls;
* Multiparametric MRI;
* EndoPAT testing;
* 6 minute walk test;
* 12-lead ECG;
* Randomization;
* Dispense study medication and issue patient diary; and
* Urine sample collection.

At this visit, participants will be randomized to receive either liraglutide or pioglitazone first. Participants that are already taking certain classes of glucose-lowering medications may be excluded from the study (see exclusion criteria for more detail). Participants will continue to take their previously prescribed medications throughout the study.

After 16 weeks of treatment (Visit 2), participants will return to the research centre and have the following assessments:

* Vital signs;
* Physical examination;
* Blood pressure;
* Weight;
* Venepuncture (fasting sample): 20mls;
* 12-lead ECG;
* Multiparametric MRI;
* EndoPAT testing;
* 6 minute walk test;
* Check current medication list and patient clinical status;
* Check study medication compliance (diary review); and
* Urine sample collection.

Participants will then have an 8 week washout period, in which they will take no study drug. After these 8 weeks, they will return to the research centre (Visit 3) and have the same assessments as listed above for Visit 2. They will start taking the second study drug for 16 weeks.

After 16 weeks, participants will attend the research centre for a final time (Visit 4) and have the same assessments as listed above for Visit 2.

Multiparametric MRI assessments will consists of 2 parts: Magnetic Resonance Spectroscopy (MRS): The relative concentration of phosphocreatine to ATP (PCr/ATP) by 31P-MRS and cardiac and hepatic triglyceride content by 1H-MRS.

Collected blood will be tested for triglycerides, alanine aminotransferase, haemoglobin, haematocrit, creatinine, estimated glomerular filtration rate, N-terminal pro-B-type natriuretic peptide, insulin, free fatty acids, adiponectin, glucose and lipid profiles, glutamic acid decarboxylase antibodies, and Zinc transporter 8 antibodies. Urine will be spot-tested for albumin/ creatinine ratio.

Previous clinical studies have found an association between diabetes and impaired function of the endothelium of blood vessels. The EndoPAT 2000 is a machine that measures endothelium function via 2 thimble-sized sensors placed on the index fingers. This is a safe and non-invasive way of testing the condition of the participant's blood vessels, and testing takes about 5 minutes.

The 6 minute walk test is an exercise test that requires patients to walk along a long flat corridor for 6 minutes to see how far they can walk at their own pace.

Liraglutide will be administered at 0.6mg once daily to start, then titrated up to 1.2mg after 2 weeks if the participant's glucose levels permit. Participants will be trained how to administer the injection themselves. Glucose assessments will be done after 2 weeks of treatment with Liraglutide. Pioglitazone is taken orally. Participants will be started on 15mg once daily; this will be titrated up to 30mg after 2 weeks then to 45mg after another 2 weeks if glucose levels permit. Glucose assessments will be done 2 weeks after starting treatment, then 4 weeks after starting treatment. Participants will be told to continue their usual schedule of glucose monitoring at home while on the study drugs (no additional monitoring at home will be necessary).

Participants will be given diaries to complete while they are on both drugs.

ELIGIBILITY:
Inclusion Criteria:

Lean cohort

1. Men and women>18 years of age;
2. Normal body weight (18.5 ≤ BMI ≤25 kg/m2);
3. T2D patients can be on treatment with oral glucose lowering therapies, and if they are, they must have been on these treatments for at least 12 weeks prior to screening;
4. 6.5≤HBA1c≤10% at screening;
5. Agreement to maintain prior diet and exercise habits for the duration of the study.

Overweight cohort

1. Men and women>18 years of age;
2. Increased body weight (BMI >27 kg/m2);
3. T2D patients can be on treatment with oral glucose lowering therapies, and must have been on these treatments for at least 12 weeks prior to screening;
4. 6.5≤HBA1c≤10% at screening;
5. Agreement to maintain prior diet and exercise habits for the duration of the study.

Exclusion Criteria:

1. Any type of diabetes other than T2D;
2. Past history of significant CAD;
3. Known HF;
4. Significant renal impairment (eGFR<30ml/min/m2);
5. Participation in a clinical trial of an investigational medicinal product (CTIMP) in the preceding 12 weeks;
6. Known hypersensitivity to dobutamine or gadolinium or any other contra-indications to MRI;
7. Participants with obesity where their girth exceeds the scanner bore;
8. History of pancreatitis;
9. Any history of liver disease;
10. Patients with Multiple Endocrine Neoplasia syndrome type 2 (MEN 2);
11. Prior or current use of thiazolidinediones (aka PPAR-γ agonists), fibrates, GLP-1RA or insulin;
12. Patients that are pregnant (female participants only);
13. Inflammatory bowel disease
14. Diabetic gastroparesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in myocardial perfusion after treatment | 40 weeks
  Measured changes in myocardial perfusion by Magnetic Resonance Imaging (MRI) after treatment with liraglutide and pioglitazone.

SECONDARY OUTCOMES:
Myocardial energetics (PCr/ATP ratio) | 40 weeks
  Change in myocardial energetics as measured by MRI after treatment
Myocardial steatosis (myocardial triglyceride content) | 40 weeks
  Change in myocardial steatosis as measured by MRI after treatment
Myocardial function | 40 weeks
  Change in myocardial function as measured by MRI after treatment
Insulin resistance (HOMA-IR) | 40 weeks
  Change in HOMA-IR as determined by blood results after treatment
Physical performance | 40 weeks
  Change in physical performance as measured by 6 minute walk test after treatment
Hepatic steatosis (hepatic triglyceride content) | 40 weeks
  Change in hepatic steatosis as measured by MRI after treatment
Peripheral endothelial function | 40 weeks
  Changes in peripheral endothelial function as measured by EndoPAT after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals Trust, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Derived] Chowdhary A, Thirunavukarasu S, Joseph T, Jex N, Kotha S, Giannoudi M, Procter H, Cash L, Akkaya S, Broadbent D, Xue H, Swoboda P, Valkovic L, Kellman P, Plein S, Rider OJ, Neubauer S, Greenwood JP, Levelt E. Liraglutide Improves Myocardial Perfusion and Energetics and Exercise Tolerance in Patients With Type 2 Diabetes. J Am Coll Cardiol. 2024 Aug 6;84(6):540-557. doi: 10.1016/j.jacc.2024.04.064. PMID 39084829